CLINICAL TRIAL: NCT04993222
Title: A Randomized, Open-label, Two-preparation, Single-dose, Two-sequence Pilot Bioequivalence Study Between Amphotericin B Liposome for Injection and AmBisome® in Healthy Subjects
Brief Title: A Pilot Bioequivalence Study Between Amphotericin B Liposome for Injection and AmBisome® in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HC1507YBE201901
Record Dates: First submitted 2021-07-07; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Amphotericin B; Injections; liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence TR (Experimental): 6 healthy subjects assigned to the sequence TR were administrated intravenously for 120 mins with the test product of amphotericin B liposome for injection in period 1 and the reference product of AmBisome® in period 2.
  Interventions: Drug: Amphotericin B liposome for injection; Drug: AmBisome®
- Sequence RT (Experimental): 6 healthy subjects assigned to the sequence RT were administrated intravenously for 120 mins with the reference product of AmBisome® in period 1 and the test product of amphotericin B liposome for injection in period 2.
  Interventions: Drug: Amphotericin B liposome for injection; Drug: AmBisome®

INTERVENTIONS:
Drug: Amphotericin B liposome for injection — IV infusion
  Other Names: the test product
Drug: AmBisome® — IV infusion
  Other Names: the reference product

SUMMARY:
The 2 × 2 crossover designed study is to evaluate the bioequivalence of two different amphotericin B liposome for injection after single IV infusion at the same dose in normal healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign informed consent.
2. Healthy female and male volunteers aged 18-55 years.
3. Body weight ≥ 50 kg for male and ≥ 45 kg for female with a body mass index (BMI) in the range of 19.0 to 26.0 kg/m2 (inclusive).
4. Subjects must be in good health on the basis of medical history, physical examination, electrocardiogram, chest X-ray, and routine laboratory evaluations.
5. Able to communicate well with the investigator and comply with the requirements of the study.

Exclusion Criteria:

1. History of allergic reactions to amphotericin B or its analogs. History of allergy to two or more kinds of drugs or food.
2. Subjects have any history of surgery, trauma that may affect the safety of the study or the intracorporal process of the drug, or have a surgical schedule during the study period.
3. Use of any prescription or over the counter medication within 14 days prior to screening.
4. History of drug abuse within 6 months prior to screening.
5. Smoking more than 5 cigarettes per day within 3 months prior to screening, or unable to stop using any tobacco products during the trial period.
6. Consumption of alcohol in excess of 14 units/week within 3 months prior to screening.
7. Consumption excessive amounts of tea, coffee and/or caffeine-rich beverages daily within 3 months prior to screening.
8. Participation in other trial within 3 months prior to screening.
9. Donation or loss of more than 400 mL blood within 3 months prior to screening.
10. Subject (female) is lactating or pregnant.
11. Subject who cannot tolerate venipuncture or have a history of needle and blood sickness.
12. Subject who has special requirements on diet and cannot accept the uniform diet.
13. Subject who has childbearing plan, unwillingness or inability to use effective contraceptives from 2 weeks before the screening to 6 months after the last dosing of the study drug.
14. Any positive test result for Hepatitis B surface antigen, hepatitis C virus antibody, anti-human immunodeficiency virus antibody or anti-syphilis spirochete.
15. Female subjects with positive pregnancy test results during the screening period or during the study.
16. Positive test result for alcohol screening or drug abuse.
17. AST or ALT, total or direct bilirubin, alkaline phosphatase and creatinine are above the upper limit of normal and potassium is below the lower limit of normal; any other abnormalities in laboratory tests and ancillary tests that are judged by the investigator to be clinically significant.
18. Not suitable for this study as determined by the investigator due to other reasons.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax | predose, 0.5, 1.0, 1.5, 2.0,2.25,2.5,3.0,4.0,6.0,8.0,10.0,14.0,26.0,50.0,74.0,146,218,290,362,434,506,578,674 hours after intravenous infusion
  90% CI of Cmax of liposome-encapsulated and non-liposome-encapsulated Amphotericin B between Amphotericin B liposome for injection and AmBisome® within 80.00%~125.00%.
Bioequivalence based on AUC0-t | predose, 0.5, 1.0, 1.5, 2.0,2.25,2.5,3.0,4.0,6.0,8.0,10.0,14.0,26.0,50.0,74.0,146,218,290,362,434,506,578,674 hours after intravenous infusion
  90% CI of AUC0-t of liposome-encapsulated andnon-liposome-encapsulated Amphotericin B between Amphotericin B liposome for injection and AmBisome® within 80.00%~125.00%.
Bioequivalence based on AUCinf | predose, 0.5, 1.0, 1.5, 2.0,2.25,2.5,3.0,4.0,6.0,8.0,10.0,14.0,26.0,50.0,74.0,146,218,290,362,434,506,578,674 hours after intravenous infusion
  90% CI of AUC0-∞ of liposome-encapsulated and non-liposome-encapsulated Amphotericin B between Amphotericin B liposome for injection and AmBisome® within 80.00%~125.00%.

SECONDARY OUTCOMES:
Tmax of liposome-encapsulated and non-liposome-encapsulated Amphotericin B | predose, 0.5, 1.0, 1.5, 2.0,2.25,2.5,3.0,4.0,6.0,8.0,10.0,14.0,26.0,50.0,74.0,146,218,290,362,434,506,578,674 hours after intravenous infusion
  Time of maximum observed concentration
t1/2 of liposome-encapsulated and non-liposome-encapsulated Amphotericin B | predose, 0.5, 1.0, 1.5, 2.0,2.25,2.5,3.0,4.0,6.0,8.0,10.0,14.0,26.0,50.0,74.0,146,218,290,362,434,506,578,674 hours after intravenous infusion
  Terminal elimination half-life
λz of liposome-encapsulated and non-liposome-encapsulated Amphotericin B | predose, 0.5, 1.0, 1.5, 2.0,2.25,2.5,3.0,4.0,6.0,8.0,10.0,14.0,26.0,50.0,74.0,146,218,290,362,434,506,578,674 hours after intravenous infusion
  Apparent elimination rate constant
Residual area of liposome-encapsulated and non-liposome-encapsulated Amphotericin B | predose, 0.5, 1.0, 1.5, 2.0,2.25,2.5,3.0,4.0,6.0,8.0,10.0,14.0,26.0,50.0,74.0,146,218,290,362,434,506,578,674 hours after intravenous infusion
  Extrapolated area
Number of treatment-emergent adverse events for the test and the reference products | predose, 0.5, 1.0, 1.5, 2.0,2.25,2.5,3.0,4.0,6.0,8.0,10.0,14.0,26.0,50.0,74.0,146,218,290,362,434,506,578,674 hours after intravenous infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Medical Treatment Center, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No